CLINICAL TRIAL: NCT06020612
Title: Desmoplasia in Cutaneous Squamous Cell Carcinoma: Inter Observer Agreement Between Dermatopathologists.
Brief Title: Interobserver Variability Desmoplasia
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-3752
Record Dates: First submitted 2023-08-18; First posted 2023-08-31 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Cutaneous Squamous Cell Carcinoma; Pathology; Recurrence; Metastasis
Keywords: Interobserver variability; Interobserver agreement; Reproducibility; Dermatopathologist; Desmoplasia
MeSH Terms: conditions — Recurrence; Neoplasm Metastasis; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Presence of desmoplasia: Tumors with presence of desmoplasia according to the predefined definition.
  Interventions: Other: Assessment by dermatopathologists
- Absence of desmoplasia: Tumors in absence of desmoplasia according to the predefined definition.
  Interventions: Other: Assessment by dermatopathologists

INTERVENTIONS:
Other: Assessment by dermatopathologists — Histological assessment of the cSCCs by eight dermatopathologists.

SUMMARY:
According to the most recent guideline of the National Comprehensive Cancer Network (NCCN), desmoplasia is considered to be a very high risk factor for recurrence, metastasis and death in cutaneous squamous cell carcinoma (cSCC). The presence of desmoplasia is assessed by dermatopathologists during histological examination of cSCCs. However, the inter-observer agreement is between dermatopathologists in the assessment of desmoplasia is unclear. Studies on inter-observer variability in the assessment of differentiation grade in cSCCs showed that there is only a weak to moderate agreement among dermatopathologists in the assessment of differentiation grade (2-4). This study aims to investigate the interobserver agreement of desmoplasia between dermatopathologists. In this prospective study, 50 cSCCs will be assessed for desmoplasia by at least eight dermatopathologists using a predefined definition.

ELIGIBILITY:
Inclusion Criteria:

* Histological coupes of patients with a cSCC between 2010 and 2018 (both cSCC with and without desmoplasia are included)
* Treated at the Maastricht University Medical Center+ (MUMC+)in Maastricht for their cSCC
* Of which the histology is available in the MUMC+

Exclusion Criteria:

- None

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of adult patients, both male and female, who were treated at MUMC+ between 2010 and 2018 for a cSCC, with and without desmoplasia, and whose histology is available.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Interobserver agreement | Through study completion, an average of 2 months
  Interobserver agreement between dermatopathologists in the assessment of desmoplasia, expressed as percentages and Fleiss' kappa (Landis and Koch, see below) <0 Poor agreement 0.0-0.20 Slight agreement 0.21-0.40 Fair agreement 0.41-0.60 Moderate agreement 0.61-0.80 Substantial agreement 0.81-1.00 Almost perfect agreement

SECONDARY OUTCOMES:
Definitions used | Before the histological assessment, at baseline.
  A description of the different definitions of desmoplasia used by the dermatopathologists.

CONTACTS AND LOCATIONS:
Overall Officials: K Mosterd, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center+, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] National Comprehensive Cancer Network. Squamous Cell Skin Cancer (Version 2.2022) May 2, 2022. Retrieved from https://www.nccn.org/professionals/physician_gls/pdf/squamous.pdf
- [Background] Prezzano JC, Scott GA, Lambert Smith F, Mannava KA, Ibrahim SF. Concordance of Squamous Cell Carcinoma Histologic Grading Among Dermatopathologists and Mohs Surgeons. Dermatol Surg. 2021 Nov 1;47(11):1433-1437. doi: 10.1097/DSS.0000000000003213. PMID 34482328
- [Background] Fujimoto M, Yamamoto Y, Takai T, Fujimoto N, Ogawa K, Yoshikawa T, Matsuzaki I, Takahashi Y, Iwahashi Y, Warigaya K, Kojima F, Jinnin M, Murata SI. Tumor Budding Is an Objective High-risk Factor Associated With Metastasis and Poor Clinical Prognosis in Cutaneous Squamous Cell Carcinoma Sized <4 cm. Am J Surg Pathol. 2019 Jul;43(7):975-983. doi: 10.1097/PAS.0000000000001284. PMID 31094931
- [Background] Nash J, Shahwan KT, Chung C, Abidi N, Gokun Y, Pan X, Carr DR. Grading of differentiation in cutaneous squamous cell carcinoma: Evaluation of interrater and intrarater reliability. J Am Acad Dermatol. 2022 Oct;87(4):895-897. doi: 10.1016/j.jaad.2021.12.015. Epub 2021 Dec 15. No abstract available. PMID 34920027
- [Background] Landis JR, Koch GG. The measurement of observer agreement for categorical data. Biometrics. 1977 Mar;33(1):159-74. PMID 843571